CLINICAL TRIAL: NCT02308904
Title: Reproductive Capacity and Association to Iron Burden and Chelation Patterns in Thalassemia Major Patients
Brief Title: Reproductive Capacity and Iron Burden in Thalassemia
Acronym: Fertility thal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CICL670AUS46T
Record Dates: First submitted 2014-11-25; First posted 2014-12-04 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: THALASSEMIA MAJOR
Keywords: Infertility; Thalassemia; Iron overload; Pituitary Iron Load; Oxidative Stress; REPRODUCTIVE CAPACITY AND ASSOCIATION TO IRON BURDEN AND CHELATION PATTERNS IN THALASSEMIA MAJOR PATIENTS
MeSH Terms: conditions — beta-Thalassemia; Infertility; Thalassemia; Iron Overload | interventions — Mass Screening; Biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Laboratory Studies for Pituitary-Gonadal Function (Other): Females: We expect to enroll approximately 15 females ages 12 years and older.
  Males: We expect to enroll approximately 15 males ages 12 years and older.
  Interventions: Other: Blood Draw/Semen Exam
- Data on iron burden and chelation history (Other): Retrospective data, as listed in this section, will be obtained from chart review and results of relevant clinical data.
  1. Iron burden data
  2. Assay for non-transferrin bound iron (NTBI)
  3. Chelation data
  4. Oxidant stress
  5. History or presence of hypogonadism
  Interventions: Other: Retrospective data/Chart Review/Relevant Clinical Results
- Pituitary MRI (Other): MRI has been shown to demonstrate well the changes related to iron toxicity in the pituitary gland.
  Interventions: Other: Pituitary MRI

INTERVENTIONS:
Other: Blood Draw/Semen Exam — Females:
  1. Obtain levels of LH/FSH, Estradiol, and AMH in all enrolled women. Males: We expect to enroll approximately 15 males ages 12 years and older.
  1. Levels of FSH/LH and testosterone will be obtained. In addition, we will examine the association of the hormone inhibin B with mean fertility measures. Inhibin B levels were shown to correlate with azospermia and could demonstrate better prediction of reproductive potential.
  2. Semen exam for determination of volume, sperm count, motility and sperm DNA integrity will be determined for interested adult thalassemia males (age ≥18 years and older).
  Other Names: Screening for biomarkers and correlations with iron load
  Arms: Laboratory Studies for Pituitary-Gonadal Function
Other: Retrospective data/Chart Review/Relevant Clinical Results — 1. 1. Documentation of liver iron from SQUID or MRI. 2. Transfusion data on age at onset of regular transfusions, transfusion frequency over the previous five years, and years of chronic transfusion therapy (defined as 8 or more per year). 3. Data on cardiac iron as indicated by T2* MRI. 4. Ferritin levels.
  2. NTBI will be accessed using a mobilizer ligand to collect NTBI from all pools as Fe-NTA which is then measured by HPLC.
  3. 1. Age at onset of chelation 2. Estimated periods of known or recalled non-compliance with regular chelation. 3. Listing of all chelation drugs previously used including dose and time period.
  4. 1. Vitamins E and C, at time closest to obtaining reproductive hormone levels. 2. Measuring the ratio of reduced gluthatione (GSH) to oxidized gluthatione (GSSG).
  5. Assessment of time for pubertal development, assessment of menstrual history and need for treatment with gonadal hormone replacement.
  Arms: Data on iron burden and chelation history
Other: Pituitary MRI — MRI has been shown to demonstrate well the changes related to iron toxicity in the pituitary gland. An MRI protocol was optimized at Children's Hospital and Research Center Oakland (CHRCO) and Texas Children's Hospital. Utilizing 1.5 T clinical scanner to evaluate the iron accumulation in the anterior pituitary. The total data acquisition time is approximately 32 minutes. No sedation will be given.
  MRI data will be sent to Dr. Wang, department of Radiology, Children's Medical Center, University of Texas Southwestern Medical Center, Dallas, Texas. Quantification of R2, pituitary height and volume will be conducted.
  Arms: Pituitary MRI

SUMMARY:
The improved long-term survival of thalassemia major (TM) patients has resulted in increased focus on the ability to preserve fertility. While the association of iron toxicity with vital organ dysfunction, heart and liver, has been extensively investigated, the correlation of reproductive capacity and extent of iron overload is not well understood. Despite remarkable progress in methodology for prediction of reproductive status and intervention for preserving fertility, implementation in thalassemia is lacking.

The investigators hypothesize that iron toxicity to the anterior pituitary occurring in the process of transfusional iron loading is directly associated with a decline in gonadal function. The investigators expect pituitary MRI measurements of iron deposition as well as markers of oxidative damage to correlate with the functional studies of pituitary-gonadal axis performed in this study. This cross sectional study will examine the relation of pituitary iron deposition and pituitary volume; serum iron and oxidative stress measures, liver iron concentration (LIC), cardiac iron and chelation adequacy with pituitary and gonadal reproductive hormone levels (and spermatogenesis in adult male patients), in order to better define the association of iron burden and chelation patterns with fertility potential, in thalassemia patients with iron overload. The study will assess whether the current chelation treatment regimens, in particular during the pubertal developmental age, are adequate for preserving fertility and could lead to improved chelation routines for preventing the high prevalence of compromised fertility. In addition, by utilizing state-of-the-art markers for fertility status, findings from this study may improve current methods for screening for hypogonadism and reproductive potential and allow earlier intervention.

The investigators propose to examine 26-30 patients, 12 years and older, with measures of fertility potential, and correlate them to their current iron burden parameters and to the cumulative iron effect as indicated by past iron overload patterns and chelation history.

ELIGIBILITY:
Inclusion Criteria:

* Transfusion-dependent* females and males with thalassemia (any genotype) who are 12 to 45 years of age.
* History of at least 5 years of chronic transfusion (defined as ≥ 8 transfusions/year) (Age of initiation of transfusions does not matter)
* Any pubertal stage.
* Liver iron evaluated by SQUID, MRI or liver biopsy within 12 months prior to enrollment in the study.
* Need to be able to stop hormonal therapy for 3 weeks (males) and one month (females) prior to study enrollment.

Exclusion Criteria:

* Pregnant or lactating during study enrollment
* Unable to obtain liver iron concentration within 12 months prior or 6 months after study entry.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Laboratory studies for pituitary and gonadal function and for iron level measures | Up to 12 months
  Each patient's pituitary iron and pituitary volume will be correlated with each hormone levels: LH, FSH, estrogen and AMH (Females), testosterone Inhibin B and (males).
  We will then evaluate potential associations using Pearson correlations. Univariate analyses on all variables and it's relation with iron, will also be conducted.

SECONDARY OUTCOMES:
Retrospective analysis of annual LIC and of type and dose of iron chelation agent in the parallel time period | Up to 12 months
  We will evaluate potential associations using Pearson correlations of each measure: Mean LIC with each of the fertility hormone levels and with pituitary volume and height. Mean ferritin with each of the fertility hormone levels and with pituitary volume and height. NTBI with each of the fertility hormone levels and with pituitary volume and height. Oxidative measures (Vit C, Vit E, GSH/GSSG) with each of the fertility hormone levels and with pituitary volume and height. Regression analysis will be utilized to assess correlation of pituitary iron, LIC and cardiac iron. We will compute descriptive statistics for all measures by group. We will assess differences between the 2 groups using Student's t-test for continuous data and chi-square or Fisher's exact for categorical. A detailed retrospective analysis of LIC and chelation patterns (type of chelator and average dose) on these 2 groups will also be performed and fertility measures will be compared.

OTHER OUTCOMES:
Pituitary MRI and Male: Semen analysis | Up to 12 months
  Pituitary iron and pituitary volume will be correlated with sperm count and with DNA breakage in males (≥18 years old) who have these test results. Statistical methods as detailed under primary objective, will be utilized.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia T Singer, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- UCSF Benioff Children's Hospital Oakland, Oakland, California, United States